CLINICAL TRIAL: NCT04089163
Title: Toca 8: A Multicenter, Open-Label, Phase 1 Study to Evaluate the Safety and Tolerability of Toca 511, a Retroviral Replicating Vector, Combined With Toca FC in Patients With Recurrent High Grade Non-Muscle Invasive Bladder Cancer
Brief Title: A Study of Toca 511 & Toca FC in Patients With Recurrent High Grade Non-Muscle Invasive Bladder Cancer (Toca 8)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-19-01
Record Dates: First submitted 2019-08-30; First posted 2019-09-13 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Bladder Cancer
Keywords: non-muscle invasive bladder cancer; bladder cancer; high grade non-muscle invasive bladder cancer; HG NMIBC; NMIBC; high grade NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — vocimagene amiretrorepvec; Flucytosine

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design with expansion at recommended Phase 2 dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential Dose Cohorts (Experimental): Doses of Toca 511 will be evaluated in sequential cohorts. Toca 511 will be administered as a single intravesical instillation. Following Toca 511 administration, Toca FC will be administered orally at a dose of 220 mg/kg/day for 7 days every 6 weeks.
  Interventions: Biological: Toca 511; Drug: Toca FC (extended-release formulation of flucytosine)

INTERVENTIONS:
Biological: Toca 511 — Toca 511 consists of a purified retroviral replicating vector encoding a modified yeast cytosine deaminase (CD) gene. The CD gene converts the antifungal drug, flucytosine (5-fluorocytosine; 5-FC) to the anticancer drug 5-fluorouracil (5-FU) in cancer cells that have been infected by the Toca 511 vector.
  Other Names: vocimagene amiretrorepvec; retroviral replicating vector (RRV)
Drug: Toca FC (extended-release formulation of flucytosine) — Toca FC is an extended-release formulation of flucytosine and is supplied as 500 mg tablets
  Other Names: flucytosine; 5-fluorocytosine (5-FC)

SUMMARY:
This is a Phase 1, multicenter, open-label study of intravesical Toca 511 followed by oral Toca FC in patients with high grade (HG) non-muscle invasive bladder cancer (NMIBC), with cohort expansion at the recommended Phase 2 dose. Patients with recurrent HG NMIBC who are undergoing planned transurethral resection of bladder tumor (TURBT) will be enrolled into the study, subject to meeting all entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate
* At least 18 years of age
* Recurrent HG NMIBC, with HG tumor on previous histopathology
* Undergoing planned TURBT and biopsy of CIS suspicious areas
* No imaging findings consistent with T2 or greater disease, hydronephrosis, extravesical disease, nodal involvement, metastases, or other malignancies.
* Able and willing to wait at least 2 weeks following intravesical administration of Toca 511 to undergo TURBT
* If patient is a candidate for standard of care (SOC) intravesical therapy, able and willing to wait at least 2 weeks post-TURBT for initiation of such treatment
* Patient is able to be catheterized and is anticipated to be able to retain Toca 511 for approximately 2 hours
* Estimated life expectancy of at least 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Patient has adequate organ function, as indicated by the following laboratory values

  * Complete blood count: hemoglobin ≥ 10 g/dL, platelet count ≥ 100,000/mm^3, absolute neutrophil count ≥ 1,500/ mm^3, absolute lymphocyte count ≥ 500/ mm^3
  * Liver: total bilirubin ≤ 1.5 × the upper limit of normal (ULN; unless known Gilbert's syndrome); alanine aminotransferase ≤ 2.5 × ULN
  * Kidney: estimated glomerular filtration rate (GFR: Cockcroft-Gault) ≥ 50 mL/min
* Women of childbearing potential (defined as not postmenopausal [ie, ≥ 12 months of non-therapy-induced amenorrhea] or not surgically sterile) must have a negative serum pregnancy test within 7 days prior to administration of Toca 511, and be willing to use an effective means of contraception in addition to barrier methods (condoms) for the duration of the study.
* Patient and partner are willing to use condoms for 12 months after receiving Toca 511 and/or 30 days after the last dose of Toca FC, and/or until there is no evidence of the virus in his/her blood or urine, whichever is longer.

Exclusion Criteria:

* History of urothelial cancer in the upper tract or urethra; muscle invasive bladder cancer; or metastatic bladder cancer
* History of bladder tumors other than urothelial carcinoma (ie, neuroendocrine, adenocarcinoma, or squamous cell carcinoma)
* Treatment with intravesical agents within 28 days prior to Toca 511 administration
* TURBT within 12 weeks prior to planned Toca 511 administration
* History of pelvic radiation
* Bladder tumor located within a bladder diverticulum
* Genitourinary procedures (eg, prostate surgery; treatment of ureteral stones or moderate to extensive urethral stricture disease) prior to, during, or planned within the 4 weeks following TURBT, other than procedures for treatment of bladder tumors
* Severe lower urinary tract dysfunction clinically manifest as poor capacity, disabling incontinence, chronic catheter use, or chronic infections or stones
* Presence of suprapubic catheter
* History of other malignancy, unless the patient has been disease-free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as cervical carcinoma in situ or localized prostate carcinoma, after curative treatment. (Note: Men with very low or low risk prostate cancer on active surveillance are acceptable candidates for this study.)
* Active infection requiring antibiotic, antifungal, or antiviral therapy within 2 weeks prior to administration of Toca 511
* Investigational treatment within 2 weeks or immunotherapy or antibody therapy within 28 days prior to Toca 511 administration, and/or has not recovered from toxicities associated with such treatment
* Chronic treatment with autoimmune medications
* Human immunodeficiency virus (HIV) seropositive
* Pregnant or breast feeding
* Bleeding diathesis, or required to take anticoagulants or antiplatelet agents, including nonsteroidal anti-inflammatory drugs, that cannot be stopped for surgery
* Severe pulmonary, cardiac, or other systemic disease, specifically:

  * New York Heart Association > Class II congestive heart failure that is not controlled on standard therapy within 6 months prior to Toca 511 administration
  * Uncontrolled or significant cardiovascular disease, clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes), clinically significant pulmonary disease (such as ≥ Grade 2 dyspnea)
  * Any other serious medical, social, or psychological condition that, based on Investigator assessment, may affect the patient's compliance or place the patient at an increased risk of potential treatment complications
* History of allergy or intolerance to flucytosine
* Presence of a condition that would prevent the patient from being able to swallow Toca FC tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 5 weeks
  * Any treatment-related Grade 3 or higher non-hematologic toxicity, excluding nausea, vomiting, or diarrhea that are controllable with appropriate medical measures (eg, antiemetics, antimotility drugs)
  * Any treatment-related Grade 4 or higher hematologic toxicity

SECONDARY OUTCOMES:
Differences in viral transduction of Toca 511 at each dose level, based on quantitation of viral RNA and DNA in tumor | 3 weeks (+/- 1 week)
Clearance of viral RNA in plasma and urine, based on real-time quantitative reverse transcription polymerase chain reaction (qRT-PCR), and of viral DNA in whole blood and urine, based on quantitative PCR (qPCR) | 1 week for plasma, 4 weeks for urine

OTHER OUTCOMES:
Changes from baseline in immune activity in tumor, peripheral blood, and urine | 21 weeks
Complete response rate at 6 and 12 months in patients with carcinoma in situ (CIS) | Proportion of patients with CIS with complete response at 6 and 12 months
High-grade recurrence-free survival | Event free survival overall and at 6 and 12 months
Incidence of cystectomy | The proportion of patients who undergo cystectomy
Incidence of disease progression at 6 and 12 months | The proportion of patients with disease progression at 6 and 12 months

IPD SHARING:
Plan to Share IPD: No